CLINICAL TRIAL: NCT07163507
Title: Immune Response Under Immunotherapy in Lung Cancer: Study of Sputum Samples
Acronym: RICEPS-2
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: DR250196
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer (NSCLC); Lung Cancer (Non-Small Cell)
Keywords: immunotherapy; sputum samples
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — sputum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lung cancer is the leading cause of cancer-related death worldwide, with nearly 2.48 million cases and 1.8 million deaths in 2022. Despite therapeutic progress, late diagnosis and high mortality make it a major public health issue. Immune checkpoint inhibitors (ICI) such as nivolumab, pembrolizumab, and atezolizumab have improved outcomes for some patients, but only a small proportion benefit, and side effects can be severe. Research is focusing on combining ICIs with chemotherapy, radiotherapy, or other immunotherapies, but reliable biomarkers to predict responders are still lacking. The tumor microenvironment, which promotes resistance, is a promising therapeutic target. The RICEPS study (2021-2023) found specific immune cells and cytokines linked to treatment response, and the ongoing RICEPS-2 trial aims to confirm these findings in a larger group to better understand immune dynamics in lung cancer under ICI therapy.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer-related death in France and worldwide. In 2022, it affected nearly 2.48 million people and caused 1.8 million deaths. Despite therapeutic advances, it remains a major public health issue due to often late diagnosis and a high mortality rate. Over the past decade, the discovery of immune checkpoints has revolutionized treatments, particularly with the emergence of therapeutic antibodies (Abs) targeting PD-1 and PD-L1 proteins, such as nivolumab, pembrolizumab, and atezolizumab. These immune checkpoint inhibitors (ICIs) have improved the management of certain patients by reactivating T lymphocytes.

Initially used in second-line metastatic non-small cell lung cancer (NSCLC), ICIs have gradually been integrated into first-line therapy and for less advanced stages. They are currently indicated as monotherapy or in combination with chemotherapy in several settings: metastatic, as post-operative adjuvant treatment, or as consolidation therapy after radio-chemotherapy. However, only a small percentage of patients actually benefit from these therapies, and their side effects can be severe.

Current research aims to improve the response to ICIs by combining them with chemotherapy, radiotherapy, or other immunotherapies targeting new checkpoints (anti-TROP2, anti-TIGIT). However, reliable clinical criteria for identifying responder patients are still lacking. PD-L1 expression appears to be a potential marker, but its efficacy remains variable across studies. Many other biomarkers have been explored, such as mutational load, tumor infiltration by T lymphocytes, or certain blood parameters, but none have yet provided reliable prediction.

The lung tumor microenvironment plays a key role in progression and treatment resistance. Composed of tumor, stromal, and immune cells, it promotes immunosuppression and limits the effectiveness of treatments by activating resistance mechanisms. It therefore represents a promising therapeutic target for improving the response to ICIs.

The RICEPS study, conducted at the Tours University Hospital and within INSERM U1100, from 2021 to 2023, analyzed the blood and pulmonary immune response in 19 patients receiving pembrolizumab, collecting blood samples and sputum. It highlighted the presence of specific non-circulating lymphocytes, resident memory T cells (RMTs), as well as key cells in the response to ICIs, CD8 T cells, in the patients' sputum, with longitudinal follow-up. Preliminary results of this study showed that CD8+ T lymphocytes, monocytes, B lymphocytes, and several cytokines (GCSF, interleukin-4 (IL-4), IL-6, IL-7, IL-12, IL-17, IL-33) influence treatment response in the blood, regardless of treatment, patient, or time. In sputum, TRM lymphocytes and two cytokines (IL-7 and CCL2) appear to contribute to treatment response.

Based on these results, the RICEPS-2 study aims to include a larger number of patients treated with immunotherapy, regardless of lung cancer type or stage. It will analyze different cell populations, including effector and TRM lymphocytes, as well as neutrophils, to better understand the involvement of the lung mucosa in the response to ICIs. Two analysis points are planned: at the start of treatment and after three months. The hypothesis tested in this project is that immune analysis at the pulmonary level could provide valuable information on the dynamic changes in innate and adaptive immune responses at the beginning of ICI treatment in lung cancer. We hypothesize that the evolution of the immune response of patients receiving ICI differs depending on whether they are responders or not to treatment. As an additional exploratory hypothesis, we wish to compare the immune profiles at the beginning of treatment, at 3 months of treatment of patients according to their response or not to immunotherapy at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older

  * Diagnosis of localized, locally advanced, or metastatic lung cancer (NSCLC or SCLC)
  * Treatment with anti-PD1 or anti-PDL1 ICI (nivolumab, pembrolizumab, atezolizumab, durvalumab, cemiplimab), with or without chemotherapy
  * First ICI injection (in a patient who has not received it before)

Exclusion Criteria:

* Patients under legal protection
* Pregnant or breastfeeding women
* Individuals who have objected to data processing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with NSCLC or SCLC treated with immune checkpoint inhibitors
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 6 months
  progression-free survival : The primary endpoint is the association of the change, between M0 and M3, in the relative frequency of cellular actors of innate and adaptive immune responses in the sputum of patients treated with ICI, with their progression-free survival (PFS) at 6 months.
Relative frequency of cellular players in innate and adaptive immune responses in the sputum of patients treated with ICI | 6 months
  The secondary endpoint is the magnitude of the association between the relative frequency of cellular players of innate and adaptive immune responses in the sputum of patients treated with ICI, with their progression-free survival (PFS) at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Marion FERREIRA, Dr, Principal Investigator — University Hospital, Tours
Locations (1):
- university hospital, Tours, Tours, France

IPD SHARING:
Plan to Share IPD: Undecided